CLINICAL TRIAL: NCT05160792
Title: Prospective Assessment to Evaluate the Comfort of GraduCheck® in Use by Healthy Volunteers
Brief Title: Comfort of GraduCheck Under Compression Bandaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Whiteley Clinic (Other)
Collaborators: Veinsense Ltd (Unknown)
Responsible Party: Principal Investigator, Mark Whiteley, Consultant Venous Surgeon, The Whiteley Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: VS-SH-2021-02
Record Dates: First submitted 2021-12-06; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Compression Bandage
Keywords: compression; bandage; wraps; pressure; ulcer
MeSH Terms: conditions — Ulcer

STUDY DESIGN:
Intervention Model Description: Single group comparison of comfort between legs - both with identical compression bandages but the index leg with a GraduCheck device under the bandage and the control leg without.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volunteers (Experimental): Index leg - compression with GraduCheck Control leg - compression without Graducheck
  Interventions: Device: Pressure monitoring system under compression bandages on index leg

INTERVENTIONS:
Device: Pressure monitoring system under compression bandages on index leg — Adding a Graducheck device under the compression bandages on the index leg and comparing to other leg, which has compression but without the device.
  Other Names: GraduCheck

SUMMARY:
The purpose of this service evaluation is to evaluate the comfort in use of GraduCheck® by volunteers, under standard compression bandages.

DETAILED DESCRIPTION:
Study Description

This is a prospective evaluation study comparing GraduCheck® under the Urgo K2 compression bandage system.

For each volunteer, the study is to be carried out over 7 days. This includes one initial visit to the clinic (The Woundcare Consultants Clinic - with a Covid-secure protocol), and the completion of an Evaluation Form at home at 24 hours, 3 days, and 7 days after the initial visit.

Those volunteers who are already on the GraduCheck® evaluation study (Prospective Assessment to Evaluate the Use of GraduCheck® in Enabling Experienced Tissue Viability Nurses to Achieve Ideal Sub-Bandage Pressures in Healthy Volunteers. IRAS: 309519) who wish to continue onto this linked study will already be in the clinic having undergone six compression system changes already, with the final compression system being one of the two involved in this study.

Volunteers should be able to remove the compression themselves at the end of the study but are welcome to return for a nurse to remove it, if preferred.

Place of study

The study is to be initiated at the Woundcare Consultants Clinic (with a Covid-secure protocol in place) on Day 0. At this venue, volunteers will be assessed, consented, randomised (if appropriate) and the Urgo K2 compression systems placed on the legs, with the GraduCheck® device on the appropriate side.

The first evaluation will be completed by the volunteer under the guidance of the TVN if needed.

The volunteer will then go home with the compression in place on both legs, the evaluation form and waterproof covers for the compression systems to allow the volunteer to have showers. The rest of the study will therefore take place at the volunteer's home.

Healthy Volunteers

Twelve (12) healthy volunteers will be recruited.

Assessment of volunteers

Before the study commences, any potential volunteer who expresses an interest in joining the study will be given a patient information sheet and a consent form.

Those that have read the patient information sheet and consent form, and still wish to be involved, will be invited in for assessment.

Healthy volunteer participants who fulfil the above criteria (part from those measured at the assessment) will be assessed to by using a Doppler Ability ultrasound device to measure the Ankle Brachial Pressure Index (ABPI), exclude any lower limb ischaemic disease. Healthy volunteer participants must have an ABPI reading between 0.8 and 1.2.

A sphygmomanometer cuff will be placed around the lower legs at the ankle, one after the other, and inflated to 40mmHg. Volunteers will need to be able to tolerate this to be included.

Consent

Healthy volunteers who fulfil the inclusion and exclusion criteria (including the assessment of ABPI and cuff inflated around the ankle), to a maximum of 12, will be invited to consent for the study.

The healthy volunteers will have been given an opportunity to discuss any points of the study or consent before signing the consent form.

As part of the consenting process, the healthy volunteers will be informed that they can withdraw at any stage, for any reason, without having to tell the organisers of their reason.

The study protocol:

Volunteers who have already completed the linked study - Prospective Assessment to Evaluate the Use of GraduCheck® in Enabling Experienced Tissue Viability Nurses to Achieve Ideal Sub-Bandage Pressures in Healthy Volunteers - IRAS: 309519 will already have the Urgo K2 compression system bandaged on one leg with the GraduCheck® device in situ.

These volunteers will only need the other leg to be bandaged by the same TVN who performed the primary leg compression, using an identical Urgo K2 dressing system, but without the GraduCheck® device in situ.

In volunteers who are taking part of this study alone, both legs will be bandaged buy a single TVN using identical Urgo K2 compression systems on each leg. The side to have the additional GraduCheck® device will be selected by envelope randomization.

The side randomised to the GraduCheck® device will be compressed first, with the TVN using the GraduCheck® results in real time to ensure optimal pressure profile. They will then repeat the same compression technique on the other leg, but without a GraduCheck® compression device being included.

The volunteer will be given 10 minutes to walk around the room or sit to get used to the compression.

They will then be asked to fill in the first evaluation sheet. This will be done in conjunction with the TVN to ensure they understand the process.

The volunteer will then be discharged home wearing the Urgo K2 compression on each leg, with the GraduCheck® device on one side. They will be discharged with the evaluation form and instructions to complete it the following day open brackets day one or close brackets day 3 and day 7.

An appointment will be made for the volunteer to return for the TVN to remove the compression and GraduCheck® device, and to hand in the completed form. if the volunteer has elected to remove the dressings themselves, they will return to hand in the GraduCheck® device and the completed evaluation form.

The process will be as follows:

A] for volunteers involved in linked study IRAS: 309519 who are continuing onto this study If the volunteer has already been involved in the study: Prospective Assessment to Evaluate the Use of GraduCheck® in Enabling Experienced Tissue Viability Nurses to Achieve Ideal Sub-Bandage Pressures in Healthy Volunteers - IRAS: 309519, this second study will continue from the end of the previous study.

By being part of the previous study, the volunteer will have already undergone assessment and will have the Urgo K2 compression system on one leg with the GraduCheck® system in place.

Therefore for these volunteers, the protocol is for the same TVN who performed their Urgo K2 compression to do the same with an identical system on the other leg.

With both legs being compressed, one with the GraduCheck® device in place, these volunteers can now join the common protocol below.

B] for volunteers new to this study

Volunteers who did not take part in the linked study Prospective Assessment to Evaluate the Use of GraduCheck® in Enabling Experienced Tissue Viability Nurses to Achieve Ideal Sub-Bandage Pressures in Healthy Volunteers - IRAS: 309519 will follow the protocol:

Each volunteer will be assessed by having their ankle brachial pressure (ABPIs) measured and noted (must be between 0.8-1.2) and have a blood pressure cuff placed around the lower leg just above the ankle on each side and inflated to 40 mm Hg to ensure they can tolerate the pressure.

Provided this assessment is satisfactory, and the inclusion/exclusion criteria are fulfilled, the volunteer will go through the consenting process for the study.

Provided that they give consent and are happy to proceed:

1. - the leg to be treated with the Urgo K2 compression system with the GraduCheck® device in place (the index leg) will be selected by envelope randomisation. It will either be left or right.
2. - the TVN will perform compression of the selected leg using the Urgo K2 as per manufacturer's instructions. However, when the first layer is put on, the GraduCheck® device will be placed on the first layer of bandaging in the anterior lateral position of the lower leg. The bandaging will then be completed using the pressure measured by the GraduCheck® device to ensure the correct pressure profile.
3. - once the compression system with GraduCheck® is in place on the index leg, the same TVN will immediately apply an identical Urgo K2 compression system to the other leg (control leg) aiming to emulate the same compression pressure that they used on the index leg.

   Common study processes
4. - the volunteer will now have an Urgo K2 compression system on both lower legs, both applied by the same TVN, with a GraduCheck® device in place on the index leg and without on the control leg.

   The volunteer will be asked to walk around and sit down as they wish to for 10 minutes.
5. - after 10 minutes, provided the volunteer is comfortable with the compression system on each leg, the volunteer will go through the Day 0 section on the evaluation form and complete it. The TVN will be present if there are any questions.
6. - the volunteer will then be allowed home with the compression system in place on both legs which will then stay in place for the next 7 days and nights (GraduCheck® k on the index side), with the evaluation form and plastic coverings for the lower legs to enable the volunteer to have showers whilst wearing the compression.
7. - the volunteer will complete the evaluation form on:

   * Day 1
   * Day 3
   * Day 7
8. - the volunteer will return to the study centre one week after the start of the study for the compression to be removed, the GraduCheck® device and evaluation form handed in. If the volunteer has removed their own compression bandaging before this time, they will bring it in to the study centre to return the compression bandaging and GraduCheck® device along with the evaluation form.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over
* Have an ankle brachial pressure index (ABPI) between 0.8-1.2 (at assessment)
* Have no active ulceration

Exclusion Criteria:

* Under the age of 18
* Unable to wear compression bandages of hosiery for any reason
* Unable to walk unaided and at normal speed for at least one mile
* Previous history of deep vein thrombosis
* Have known arterial insufficiency (an ABPI of below 0.8) (at assessment)
* Unable to tolerate a cuff at 40 mmHg around ankle (at assessment)
* Have active ulceration
* Have signs of recent lower limb trauma, active infection, ongoing untreated venous disease, or significant ankle oedema
* Unable to give informed consent
* Pregnant
* Fragile skin that may be damaged whilst trying to apply compression bandaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Comfort | 7 days
  Comfort of leg with compression and GraduCheck device compared with comfort of compression alone

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Whiteley, MS, Principal Investigator — The Whiteley Clinic Ltd

IPD SHARING:
Plan to Share IPD: No
The results will be presented at research meetings and submitted for publication in peer-reviewed journals.
  Results will be published in figures and tables and text - no data to identify individuals will be published.

REFERENCES:
- [Background] Bobbink P, Larkin PJ, Probst S. Experiences of Venous Leg Ulcer persons following an individualised nurse-led education: protocol for a qualitative study using a constructivist grounded theory approach. BMJ Open. 2020 Nov 26;10(11):e042605. doi: 10.1136/bmjopen-2020-042605. PMID 33243816
- [Background] Guest JF, Fuller GW, Vowden P. Cohort study evaluating the burden of wounds to the UK's National Health Service in 2017/2018: update from 2012/2013. BMJ Open. 2020 Dec 22;10(12):e045253. doi: 10.1136/bmjopen-2020-045253. PMID 33371051